CLINICAL TRIAL: NCT07270705
Title: Assessment of the Efficacy and Safety of OROXID® Oral Solution in Patients With Gingivitis
Acronym: OroxGing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ENIKAM d.o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OROXID-PR-03-25
Record Dates: First submitted 2025-11-19; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Gingivitis
Keywords: Gingivitis; hydrogen peroxide; mouth rinses; oral solutions
MeSH Terms: conditions — Gingivitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OROXID® forte oral solution (Experimental): Medical device: OROXID® forte oral solution
  Interventions: Device: OROXID® forte oral solution
- OROXID® sensitive oral solution (Experimental): Medical device: OROXID® sensitive oral solution
  Interventions: Device: OROXID® sensitive oral solution
- Standard of Care (Other): Oral solutions are not allowed
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: OROXID® forte oral solution — Patients will use OROXID® forte oral solution two to three times daily for 4 weeks as an adjunct to standard care.
  Arms: OROXID® forte oral solution
Device: OROXID® sensitive oral solution — Patients will use OROXID® sensitive oral solution two to three times daily for 4 weeks as an adjunct to standard care.
  Arms: OROXID® sensitive oral solution
Other: Standard of Care — Patients will receive standard of care, consisting of proper tooth brushing without the use of any mouthwash or other products intended to maintain oral hygiene or reduce oral bacterial load.
  Arms: Standard of Care

SUMMARY:
Gingivitis is a reversible inflammation of the gums caused by the accumulation of dental plaque. Without appropriate intervention-such as proper oral hygiene and plaque removal-gingivitis can progress to periodontitis, leading to clinical attachment loss, alveolar bone resorption, and ultimately tooth loss. Gingivitis can be managed with regular and proper tooth brushing and the use of interdental brushes. In cases of more extensive inflammation affecting multiple or all teeth, dental treatment may be required, including scaling, air polishing, or both. Depending on the dentist's assessment, inflamed gums may also be treated with antibiotic therapy.

As an adjunctive therapy to manage inflamed gums and maintain proper oral hygiene, the use of mouth rinses or oral solutions containing chlorhexidine, hyaluronic acid, chitosan, or active oxygen (peroxide) is recommended. These agents have antimicrobial properties, help reduce plaque accumulation, and support tissue healing. Mouth rinses containing hydrogen peroxide have been used for over a century as an adjunct to mechanical plaque removal and for the prevention or management of oral infections. Despite long-term use, clinical studies on hydrogen peroxide-based mouth rinses are limited and vary in design, which makes comparison of results difficult.

One of the objectives of the proposed post-marketing clinical study is to generate data on the safety and effectiveness of hydrogen peroxide mouth rinses as adjunctive therapy in the treatment of gingivitis. The study will evaluate two concentrations of hydrogen peroxide mouth rinses: a 1.5% solution (Oroxid® sensitive) and a 3% solution (Oroxid® forte).

ELIGIBILITY:
Inclusion Criteria:

1. Systemically healthy participants aged 18 years or older.
2. Presence of at least 20 natural teeth.
3. Probing pocket depth less than or equal to 3 mm.
4. Presence of bleeding on probing in more than 10% of sites.
5. Mean Gingival Index (Silness & Löe) of at least 1.
6. Ability and willingness to follow oral hygiene instructions after the intervention.
7. Signed informed consent form after being informed about the study.

Exclusion Criteria:

1. Periodontal treatment within the last three months.
2. Diagnosis of periodontitis.
3. Use of mouth rinses or oral gels within the last month.
4. Use of antibiotic therapy within the last three months.
5. Known allergy or hypersensitivity to any components of the investigational products.
6. Ongoing treatment with antihypertensive, antilipemic, antiarrhythmic, or other cardiovascular medications.
7. Presence of systemic diseases such as diabetes, HIV/AIDS, liver disease, chronic kidney disease, tuberculosis, or autoimmune disorders (e.g., lupus, scleroderma, Crohn's disease).
8. Use of immunosuppressive medications.
9. Ongoing orthodontic treatment, fixed orthodontic appliance, or removable denture.
10. Pregnant or breastfeeding women.
11. Smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Gingival Index (GI) at Day 7 | Baseline and Day 7
  Mean change in Gingival Index (Silness and Löe) scores from baseline to day 7, comparing the two active treatment groups (OROXID® forte and OROXID® sensitive) with the control group. The Gingival Index (GI) evaluates the severity of gingival inflammation on a scale of 0 to 3, based on redness, swelling, and bleeding on probing.
Plaque Index (PI) at Day 7 | Baseline and Day 7
  Differences in Plaque Index (PI) scores between the active and control groups will be evaluated using the Silness and Löe Plaque Index. This index assesses the thickness of dental plaque along the gingival margin based on the following scoring criteria: Score 0 = No plaque score; 1 = Mild plaque along the gingival margin; Score 2 =Moderate layer of plaque along gingival margin, interdental spaces free; Score 3 = Abundant plaque along the gingival margin, interdental spaces filled with plaque. Higher scores indicate poorer oral hygiene and greater plaque accumulation.
Bleeding on Probing (BOP) at Day 7 | Baseline and Day 7
  Difference in the presence of bleeding on probing (BOP) between the two active treatment groups and the control group after 7 days of treatment. BOP evaluates gingival inflammation by recording the presence/absence of bleeding within 30 seconds after gentle periodontal probing, serving as a key diagnostic indicator of active periodontal disease.

SECONDARY OUTCOMES:
Gingival Index (GI) at Day 14 and 28 | Baseline, Day 14, and Day 28
  Mean change in Gingival Index (Silness and Löe) scores from baseline to day 14, and 28, comparing the two active treatment groups (OROXID® forte and OROXID® sensitive) with the control group. The Gingival Index (GI) evaluates the severity of gingival inflammation on a scale of 0 to 3, based on redness, swelling, and bleeding on probing.
Plaque Index (PI) at Day 14 and 28 | Baseline, Day 14, and Day 28
  Differences in Plaque Index (PI) scores between the active and control groups will be evaluated using the Silness and Löe Plaque Index. This index assesses the thickness of dental plaque along the gingival margin based on the following scoring criteria: Score 0 = No plaque score; 1 = Mild plaque along the gingival margin; Score 2 =Moderate layer of plaque along gingival margin, interdental spaces free; Score 3 = Abundant plaque along the gingival margin, interdental spaces filled with plaque. Higher scores indicate poorer oral hygiene and greater plaque accumulation.
Bleeding on Probing (BOP) at Day 14 and 28 | Baseline, Day 14, and Day 28
  Difference in the presence of bleeding on probing (BOP) between the two active treatment groups and the control group after 14 and 28 days of treatment. BOP evaluates gingival inflammation by recording the presence/absence of bleeding within 30 seconds after gentle periodontal probing, serving as a key diagnostic indicator of active periodontal disease.
Rate of infection | Baseline to Day 28
  Incidence of infections in each group
Adverse events | Baseline to Day 28
  Number and percentage of participants experiencing adverse events (AEs) related to the use of OROXID® forte or OROXID® sensitive during the 12-week study period. The nature, severity, and relationship of each AE to the study product will be recorded and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastjan Perko, PhD, DMD, Principal Investigator — Ustna medicina d.o.o.
Locations (2):
- Slovenia (2):
  - Klinika Križaj Ljubljana, Ljubljana
  - Ustna medicina d.o.o., Ljubljana

IPD SHARING:
Plan to Share IPD: No
As a company operating under the jurisdiction of the EU, the organization is subject to the General Data Protection Regulation (GDPR), which imposes strict requirements on the processing and sharing of personal data, including health-related information. Individual Participant Data (IPD) from clinical trials is considered sensitive personal data under GDPR.Even when data is anonymized or pseudonymized, sharing IPD with third parties-especially outside the EU-requires careful assessment of data protection safeguards, appropriate legal basis, and in some cases, additional participant consent. Unless all conditions for lawful data transfer and processing are met, including compliance with GDPR Articles 44-50 concerning international data transfers, the sharing of IPD is not permitted.For this reason, and to ensure full compliance with EU data protection regulations while safeguarding the privacy and rights of study participants, individual-level data cannot currently be shared.